CLINICAL TRIAL: NCT05717075
Title: Effects of Parents Included in Decision-making During Medical Round in Neonatal Intensive Care Unit: Cross-over Randomized Controlled Trial
Brief Title: Effects of Parents Included in Medical Round of Neonatal Intensive Care Unit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nagano Children's Hospital (Other)
Responsible Party: Principal Investigator, Ryo Itoshima, Principal Investigator, Nagano Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Parents round RCT
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Family Centered Care; Decision Making
Keywords: Medical round; Doctor's round

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Parents Round, then no special round) (Other): Parents of enrolled patient receive the intervention for two weeks after the consent to the study (Period I). For two weeks after the intervention in Period I, the parents do not receive the intervention (Period II).
  Interventions: Behavioral: Parents Round
- Group B (no special round, then Parents Round) (Other): Parents of enrolled patient receive no intervention for two weeks after the consent to the study (Period I). For two weeks after Period I, the parents receive the intervention (Period II).
  Interventions: Behavioral: Parents Round

INTERVENTIONS:
Behavioral: Parents Round — The intervention carried out in this study is called Family Round. The Family Round is an additional medical round, aiming to involve parents in the discussion. The basic attitude of the healthcare staff is to make decisions collaboratively with parents or other family members based on the parents' observations of their infant and parents' opinions. As our daily medical round is carried out in the morning between 8 and 10 a.m. and we offer no accommodation for parents in the NICU, the Family Round will be carried out separately in the afternoon. One neonatologist who is in charge of the infant or taking care of the infant on that day will be a facilitator and proceed with the Parent Round according to the protocol. Other healthcare staff are also encouraged to participate, although the number of participants is limited.

SUMMARY:
The goal of this cross-over randomized controlled study is to evaluate the effects of medical rounds with parents. The main questions it aims to answer are:

* How feasible the protocol of this study is to include parents in the medical round?
* Does the Family Round promote the quality of family centered care in the NICU perceived by parents and healthcare staff?
* Does the Family Round promote parent-infant bonding?
* Does the Family Round reduce parents' anxiety?
* Does the Family Round increase parents' satisfaction?
* Does the Family Round improve staff's communication skills to integrate parents in the discussion of medical rounds?

Participants will participate in the Family Round for two weeks, which is organized by healthcare staff following a protocol aiming to integrate parents into the discussion.

They will be compared to the two-week period without the Family Round.

DETAILED DESCRIPTION:
[Intervention] The intervention included in this study is called "Parents Round," which aims to integrate parents into the discussion of medical rounds. Parents Round is organized by healthcare staff following the protocol. The protocol details are described below.

Essential requirements

* Limited number of participants: infant, parents, other important family members if present, up to 2 doctors, and up to 4 healthcare staff including doctors
* At the bedside of the infant
* All participants, excluding the infant, sit on the chair
* Privacy consideration: ask the other parents in the same room to go out or wear headphone
* Ask parents about their infant's condition and their opinion before the healthcare staff speaks
* Mention the respiration, feeding, skin-to-skin contact, and involvement in care-taking and try to make a decision collaboratively with parents about the short- or long-term plan in each item

Recommended requirements

* Quiet environment: turn off or reduce the volume of the monitor alarm
* Effective communication to promote parents' participation and involvement: parents speaking first, empathetic attitude, not interrupting while parents speak, and not frequently using the technical term, for example.
* Encourage psychologists to participate
* Nurses complement parents' role and may lead some parts of the discussion: e.g. discharge preparation

[Sample size] To detect the mean difference of 0.5 in the FCC-Q average scores (standard deviation, 0.77), with power 0.8 and alfa 0.05 in the cross-over trial, at least 40 families are necessary. We estimate the possibility of dropout as 10% and, finally, the target sample size is decided to be 46 families (or 92 parents) in total.

[Randomization] After families consent to participate, they are randomly assigned to Group A (intervention first) or Group B (no intervention first). The randomization sequence will be created using Excel 2019 (Microsoft, Redmond, WA, USA) and will be stratified based on the gestational age at birth (preterm births [born before 37 weeks of gestation] or full-term birth [born 37 weeks of gestation or later]) with a 1:1 allocation using random block sizes of 2 and 4.

The sequence allocation was conducted by a researcher in the research group who will not be involved in family enrollment. The allocated number was concealed from the researcher enrolling and assessing participating families in sequentially numbered, opaque, sealed, and stapled envelopes. This sealing will be conducted by another research member who will not be involved in the enrollment process. Black thick paper will be used inside the envelope to prevent the allocated number from being visible from the outside. The neonatologists in the study group, except for one person working outside the unit, will be responsible for the family enrollment. One of the envelopes will be opened soon after the family's consent by the person who is responsible for the enrollment according to the number written outside the envelope. To prevent subversion of the allocation sequence, the infant's name, identification number, and date of birth will be written on the envelope before opening it and on the paper on which the allocated number is printed soon after opening it. Any blinding is not possible in this study design after allocating the families.

[Statistics] The differences in each continuous outcome measures (FCC-Q, Short-STAI, and Satisfaction questionnaire) between the intervention and the control will be analyzed using the linear mixed model: including intervention/control, Period I/II, an interaction effect of the intervention and the period, and the infant's days of life at each intervention/control phase as covariates and parent as a random effect.

In addition, the proportion of parents with possible clinical state or trait anxiety will be also compared using the cutoff score of > 9.5 in state and > 13.5 in trait anxiety 8. The generalized mixed model will be used to compare the two groups: including intervention/control, Period I/II, an interaction effect of the intervention and the period, and the infant's days of life at the assessment as covariates and parent as a random effect.

The differences in the outcome measures for healthcare staff will be analyzed using the Wilcoxon rank sum test. Additionally, the adjusted outcomes will be estimated using the linear mixed model. The following variables will be included in the model: the outcome measure, occupation, and years of experience as fixed effects, and each healthcare staff as a mixed effect.

All analyses will be conducted for both parents together and individually. Separate analyses will be conducted including and excluding those who never participate in the Family Round during the study period. The differences in each question in FCC-Q or the Satisfaction questionnaire will be also compared. The state and trait anxiety measured by Short-STAI will be analyzed separately. The proportion of each rating in the Bliss Baby Charter audit tool will be compared between the groups using the Wilcoxon rank sum test. R and RStudio will be used to analyze the data. The analyses performed are two-tailed, and P <.05 is considered statistically significant.

[Data management] Running numbers will be assigned to every family after the consent. All data will be handled pseudonymously after converting the data into electronic data. Paper documents including parents' answers will be stored in a safe archive of the unit. Electronic data will be stored in a password-protected computer. All paper and electronic data will be destroyed 10 years after the final publication.

The principal investigator will be responsible for managing access to the data. The other research members will also have the right to access the digital data. The data is co-owned by the members of the research team. We do not have the plan to make the data open in the future. However, it can be shared with another personnel or research team for another scientific purpose with the permission of the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Infants in the NICU and their parents/partner
* Infants who are expected to stay in the NICU for more than one month in the future at consent

Exclusion Criteria:

no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quality of family centered care assessed by parents | 2 weeks
  The family centered care provided by the NICU is assessed by parents using FCC-Q, which was modified from DigFCC SMS questions. It consists of 9 questions: 1) active listening, 2) parent participation in infant care, 3) individualized parent education, 4) parent participation in decision-making, 5) the parental trust toward staff in infant care, 6) the parental feelings of the staff trust in infant care, 7) participation in medical round/medical care decision making, 8) received information, and 9) emotional support. The questionnaire for healthcare staff does not include question no. 7, about medical round/medical care decision making. Each question has the Likert scale from 1 to 7 (1 not at all and 7 very much; 0 if they did not visit the unit). The average score varies from 1 to 7 and a higher score indicates better family centered care received by parents.
Quality of family centered care assessed by parents | 4 weeks
  The family centered care provided by the NICU is assessed by parents using FCC-Q, which was modified from DigFCC SMS questions. It consists of 9 questions: 1) active listening, 2) parent participation in infant care, 3) individualized parent education, 4) parent participation in decision-making, 5) the parental trust toward staff in infant care, 6) the parental feelings of the staff trust in infant care, 7) participation in medical round/medical care decision making, 8) received information, and 9) emotional support. The questionnaire for healthcare staff does not include question no. 7, about medical round/medical care decision making. Each question has the Likert scale from 1 to 7 (1 not at all and 7 very much; 0 if they did not visit the unit). The average score varies from 1 to 7 and a higher score indicates better family centered care received by parents.
Quality of family centered care assessed by healthcare staff | before the enrollment of the first patient
  The family centered care provided by the NICU is assessed by parents or healthcare staff using FCC-Q, which was modified from DigFCC SMS questions. It consists of 8 questions: 1) active listening, 2) parent participation in infant care, 3) individualized parent education, 4) parent participation in decision-making, 5) the parental trust toward staff in infant care, 6) the parental feelings of the staff trust in infant care, 7) received information, and 8) emotional support. The questionnaire for healthcare staff does not include question no. 7, about medical round/medical care decision making. Each question has the Likert scale from 1 to 7 (1 not at all and 7 very much; 0 if they did not visit the unit). The average score varies from 1 to 7 and a higher score indicates better family centered care received by parents.
Quality of family centered care assessed by healthcare staff | 1 month after the end of the intervention of the last patient
  The family centered care provided by the NICU is assessed by parents or healthcare staff using FCC-Q, which was modified from DigFCC SMS questions. It consists of 8 questions: 1) active listening, 2) parent participation in infant care, 3) individualized parent education, 4) parent participation in decision-making, 5) the parental trust toward staff in infant care, 6) the parental feelings of the staff trust in infant care, 7) received information, and 8) emotional support. The questionnaire for healthcare staff does not include question no. 7, about medical round/medical care decision making. Each question has the Likert scale from 1 to 7 (1 not at all and 7 very much; 0 if they did not visit the unit). The average score varies from 1 to 7 and a higher score indicates better family centered care received by parents.

SECONDARY OUTCOMES:
Bonding feeling of parens toward their infant | 2 weeks
  The bonding feelings of parents toward their infant is assessed using the Japanese version of MIBS-J. It has ten self-report items, each of which is scored on a four-point scale (0-3). The total score varies from 0 to 30, and higher scores indicate problematic bonding feelings.
Bonding feeling of parens toward their infant | 4 weeks
  The bonding feelings of parents toward their infant is assessed using the Japanese version of MIBS-J. It has ten self-report items, each of which is scored on a four-point scale (0-3). The total score varies from 0 to 30, and higher scores indicate problematic bonding feelings.
Parents' anxiety | 2 weeks
  Parents' anxiety is assessed using the short version of the State and Trait Anxiety Inventory (Short-STAI). It was developed based on the original STAI which has 40 questions.9 The STAI assesses two different anxiety types at the same time. State anxiety is an emotional response that can change over time according to the situation. Trait anxiety indicates a personal emotional characteristic that a person has. There are 5 questions for each state and trait anxiety and each is scored on a four-point scale (1-4). The total score in each type of anxiety varies from a minimum of 5 to a maximum of 20, and higher scores indicate having more depressive symptoms.
Parents' anxiety | 4 weeks
  Parents' anxiety is assessed using the short version of the State and Trait Anxiety Inventory (Short-STAI). It was developed based on the original STAI which has 40 questions.9 The STAI assesses two different anxiety types at the same time. State anxiety is an emotional response that can change over time according to the situation. Trait anxiety indicates a personal emotional characteristic that a person has. There are 5 questions for each state and trait anxiety and each is scored on a four-point scale (1-4). The total score in each type of anxiety varies from a minimum of 5 to a maximum of 20, and higher scores indicate having more depressive symptoms.
Parents' satisfaction | 2 weeks
  Parents' satisfaction is assessed using a satisfaction questionnaire, which was made for this study purpose. It consists of 5 questions and each question is evaluated using the visual analogue scale (VAS). The VAS has a continuous bar from 0 to 100% and parents choose the point that best fits their thoughts. Here are the questions included.
  * Was the information about your baby sufficient and accurately delivered to you?
  * Did the healthcare staff listen to you well and respect your ideas?
  * When deciding how you would be involved in your baby's care, were your thoughts fully reflected?
  * When deciding your baby's future plan, were your thoughts taken into account and did you join the discussion together with the healthcare staff?
  * What is your overall level of satisfaction?
Parents' satisfaction | 4 weeks
  Parents' satisfaction is assessed using a satisfaction questionnaire, which was made for this study purpose. It consists of 5 questions and each question is evaluated using the visual analogue scale (VAS). The VAS has a continuous bar from 0 to 100% and parents choose the point that best fits their thoughts. Here are the questions included.
  * Was the information about your baby sufficient and accurately delivered to you?
  * Did the healthcare staff listen to you well and respect your ideas?
  * When deciding how you would be involved in your baby's care, were your thoughts fully reflected?
  * When deciding your baby's future plan, were your thoughts taken into account and did you join the discussion together with the healthcare staff?
  * What is your overall level of satisfaction?
Quality of medical round with parents assessed by parents | 4 weeks
  Another questionnaire will be answered by parents at the end of the study. It includes questions to explore the facilitating and inhibiting factors for parents' participation in the medical round.
Collaboration competence questionnaire of healthcare staff | before the enrollment of the first patient
  Healthcare staff's ability to work collaboratively with parents will be assessed using the collaboration competence questionnaire. The questionnaire is specifically created to assess competencies that are relevant for the Close Collaboration with Parents intervention. The questionnaire includes 21 questions that are evaluated with scale from 1 to 10 (1=not competent at all, 10=extremely competent). If the question does not ably the daily work role of the professional option "Doesn't belong to my role" can be chosen.
Collaboration competence questionnaire of healthcare staff | 1 month after the end of the intervention of the last patient
  Healthcare staff's ability to work collaboratively with parents will be assessed using the collaboration competence questionnaire. The questionnaire is specifically created to assess competencies that are relevant for the Close Collaboration with Parents intervention. The questionnaire includes 21 questions that are evaluated with scale from 1 to 10 (1=not competent at all, 10=extremely competent). If the question does not ably the daily work role of the professional option "Doesn't belong to my role" can be chosen.
Quality of family centered care assessed by healthcare staff using the Bliss Baby Charter audit tool | before the enrollment of the first patient
  The Bliss Baby Charter audit tool is a self-assessment tool to evaluate the quality of family centered care in neonatal intensive care units. The tool has 7 core principles and a total of 141 statements. All principles contain different aspects of family centered care: active care by parent and staff, parent and family support, communication, developmental care, empowered decision making, facilities, guidelines and policies, staff skills and training, information provision, and service improvement and parent involvement. Each statement is rated as green (fully delivering against all aspects of the criteria), amber (Delivering some or most of the aspects required to meet the criteria but not all), or red (Delivering none or very few of the aspects required to fulfil that criteria). The rating can be done by both healthcare staff and parents.
Quality of family centered care assessed by healthcare staff using the Bliss Baby Charter audit tool | 1 month after the end of the intervention of the last patient
  The Bliss Baby Charter audit tool is a self-assessment tool to evaluate the quality of family centered care in neonatal intensive care units. The tool has 7 core principles and a total of 141 statements. All principles contain different aspects of family centered care: active care by parent and staff, parent and family support, communication, developmental care, empowered decision making, facilities, guidelines and policies, staff skills and training, information provision, and service improvement and parent involvement. Each statement is rated as green (fully delivering against all aspects of the criteria), amber (Delivering some or most of the aspects required to meet the criteria but not all), or red (Delivering none or very few of the aspects required to fulfil that criteria). The rating can be done by both healthcare staff and parents.

CONTACTS AND LOCATIONS:
Overall Officials: +81-263-73-6700 Itoshima, MD, Principal Investigator — Nagano Children's Hospital
Locations (1):
- Nagano Children's Hospital, Azumino, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No